CLINICAL TRIAL: NCT02671110
Title: A Randomized Trial Comparing Two Approaches to Weight Loss
Brief Title: A Trial Comparing Two Approaches to Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Carels (Other)
Responsible Party: Sponsor-Investigator, Robert Carels, Professor, Bowling Green State University
Organization: Bowling Green State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 300066-10
Record Dates: First submitted 2015-11-02; First posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Overweight and Obesity
Keywords: weight loss treatment; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transforming Your Life (Experimental): The TYL program emphasized: 1) helping participants develop and maintain healthy habits and disrupt unhealthy habits, 2) enabling participants to create a personal food and exercise environment that increases exposure to healthy eating and physical activity and encourages automatic responding to goal-related cues, and 3) facilitating participants' weight loss motivation.
  Interventions: Behavioral: Transforming Your Life
- Diabetes Prevention program (Active Comparator): The DPP recommends that participants set a weight loss reduction goal of 7% or more of their baseline body weight, reduce consumption of high fat foods as a means to reduce caloric intake, and engage in brisk walking or other moderate intensity physical activity for 150 minutes per week. Sessions include information on changing energy intake and energy output through diet and exercise, and addressing psychological, social, environmental, and motivational challenges to health behavior change.
  Interventions: Behavioral: Diabetes Prevention Program

INTERVENTIONS:
Behavioral: Transforming Your Life — See Transforming Your Life Arm
  Arms: Transforming Your Life
Behavioral: Diabetes Prevention Program — See Diabetes Prevention Program Arm
  Arms: Diabetes Prevention program

SUMMARY:
This study compared the recently developed Transforming Your Life (TYL) weight loss program to the Diabetes Prevention Program (DPP), considered the "Gold Standard" in behavioral weight loss treatment.

DETAILED DESCRIPTION:
Weight loss programs evidence considerable variability in treatment outcomes and weight regain is common, signaling the need for the refinement of effective treatments. This study compared the recently developed Transforming Your Life (TYL) program to the Diabetes Prevention Program (DPP), considered the "Gold Standard" in behavioral weight loss treatment.

ELIGIBILITY:
Inclusion Criteria

1. overweight/obese (body mass index>27 kg/m2)
2. free from serious medical conditions that would complicate participation in the intervention via adherence or mobility (e.g., serious heart disease or musculoskeletal problems that would interfere with moderate exercise)
3. had not undergone bariatric surgery
4. able to provide medical clearance from their physician.

Exclusion Criteria

1. evidence of medical conditions that would complicate participation in the intervention via adherence or mobility (e.g., serious heart disease or musculoskeletal problems that would interfere with moderate exercise)
2. had undergone bariatric surgery,

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 10 months
  lbs

SECONDARY OUTCOMES:
Caloric Intake | 4 months
  kilocalories
Energy expenditure | 4 months
  kilocalories

CONTACTS AND LOCATIONS:
Locations (1):
- Bowling Green State University, Bowling Green, Ohio, United States